## The Body Project: Comparing the Effectiveness of an In-person and Virtually Delivered Intervention

NCT: 05794763

02/06/2023

Mixed effects modeling was used to control for potential lack of independence within cohort.

Specifically, for each measure we fit the following model:

$$Posttest_{ij} = \beta_0 + b_j + \beta_1 cond_{ij} + \beta_2 Pretest_{ij} + e_{ij}$$

where  $Posttest_{ij}$  is the posttest score for participant i in cohort j,  $cond_{ij}$  is an indicator variable taking on the value of 0 for control and 1 for treatment,  $Pretest_{ij}$  is the pretest score,  $b_j$  is the random intercept for cohort j, and  $e_{ij}$  is the residual. The intraclass correlation for cohort was approximately 0 for all measures, nonetheless, it was retained as this was a feature of the study design. Due to missingness at the posttest (ranged from 12% for number of eating symptoms to 24% for the other outcomes), multiple imputation was used (Graham, 2009). We imputed 50 datasets and applied Rubin's rules to pool results across the models. As a sensitivity analysis, models were fit using only participants with complete data. Models were fit in R (R Core Team, 2021) using the nlme package, the mice package was used for imputation (van Buuren, 2018) and plots were created using ggplot2 (Wickham, 2016).

## References

Graham, J.W. (2009). Missing data analysis: Making it work in the real world. *Annual Review of Psychology*, 60, 549-576.

R Core Team. (2021). *R: A language and environment for statistical computing*. (4.1) [Computer software]. R Foundation for Statistical Computing. https://www.R-project.org/.

Van Buuren, S. (2018). Flexible imputation of missing data. CRC Press.

Wickham, H. (2016). *ggplot2: Elegant Graphics for Data Analysis*. Springer Science and Business Media, LLC.